CLINICAL TRIAL: NCT02614963
Title: Effect of Clostridium Butyricum in Treating Irritable Bowel Syndrome: A Randomized, Double-blinded,Placebo- Controlled Multicenter Study
Brief Title: Effect of Clostridium Butyricum in Treating Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); Taian City Central Hospital (Other); Qingdao Eastsea Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015SDU-QILU-G13
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-03

CONDITIONS: Effect of Clostridium Butyricum in Treating Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Clostridium Butyricum
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — phosphatidyltransferase, Clostridium butyricum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clostridium Butyricum group (Experimental): Irritable bowel syndrome patients treated with Clostridium Butyricum
  Interventions: Drug: Clostridium Butyricum
- Placebo group (Placebo Comparator): Irritable bowel syndrome patients treated with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Clostridium Butyricum — Irritable bowel syndrome patients treated with Clostridium Butyricum
  Arms: Clostridium Butyricum group
Drug: placebo — Irritable bowel syndrome patients treated with placebo
  Arms: Placebo group

SUMMARY:
Clostridium Butyricum might be an effective drug in treating irritable bowel syndrome

ELIGIBILITY:
Inclusion Criteria:

* the presence of Rome III criteria for IBS ;
* Aged between 18 and 65 years old

Exclusion Criteria:

* Antibiotic, probiotic or laxative usage within 4 weeks.
* organic gastrointestinal diseases
* Severe systematic disease: diabetes mellitus, hepatic, renal or cardiac dysfunction, thyroid disease or tumor etc.
* pregnancy or lactation.
* previous major or complicated abdominal surgery.
* severe endometriosis and dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
the changes of Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) scores | 7 months

SECONDARY OUTCOMES:
IBS patients'quality of life | 7 months
  Quality of life was determined by using IBS-QOL scoring system for patients with IBS.
Composition of Microorganisms in stool | 7 months
  Primary coordination of fecal samples' 16s rDNA (ribosomal DNA) will be compared between two Groups using Braycurtis distance based Primary coordination analysis (PCoA).

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China